CLINICAL TRIAL: NCT05306015
Title: Application of Mindfulness Meditation Based on Brain Computer Interface in Radiofrequency Ablation of Atrial Fibrillation Patients
Brief Title: Application of Mindfulness Meditation Based on Brain Computer Interface in Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Zhipeng Bao
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Radiofrequency Ablation; Meditation; Pain; Fatigue; Anxiety; Depression; Brain-Computer Interfaces
MeSH Terms: conditions — Atrial Fibrillation; Pain; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Patients undergoing brain-computer interface-based mindfulness meditation training during the perioperative period of radiofrequency ablation.
  Interventions: Combination Product: Mindfulness meditation based on brain-computer interface
- control group (Active Comparator): Patients receiving routine care for radiofrequency ablation.
  Interventions: Combination Product: Routine care

INTERVENTIONS:
Combination Product: Mindfulness meditation based on brain-computer interface — Before surgery, The nurses will teach and explain the methods and significance of meditation training. Let the patient be familiar with the function and background of this method, and explain the use of the headband during the operation, so that the patient believes that meditation training can relieve pain.
  In surgery, Wear a brain-computer interface headband for the patient to collect EEG, monitor the patient's psychological changes, and provide real-time feedback.
  The patient wears a Bluetooth headset, according to the patient's preferences, different types of music are selected, and voice playback guides the patient to prepare, relax muscles and regulate breathing.
  APP judges the patient's meditation state based on EEG signals, and adjusts music, voice guidance.
  The nurse will give personalized guidance based on the patient's specific situation and the EEG displayed on the APP to help the patient achieve a state of meditation and relaxation.
  Arms: test group
Combination Product: Routine care — Give routine treatment and care, and increase or decrease the dose or adjust according to the patient's condition in accordance with the doctor's advice. Before surgery, we will introduce the level of medical care involved in the surgery and the equipment of our hospital. Inform the patient of the surgical process and possible pain, and explain in detail the cause, location and characteristics of the pain, including the time when the pain will appear and last. Instruct patients to stabilize their emotions and maintain a calm state of mind. As far as possible to meet the patient's intraoperative care needs, give psychological care, wear a headband to collect EEG signals, but do not intervene in mindfulness meditation.
  Arms: control group

SUMMARY:
In recent years, radiofrequency ablation has gradually become a first-line treatment for patients with atrial fibrillation. Radiofrequency ablation is an invasive procedure that lasts several hours, patients can experience varying degrees of discomfort and pain despite the use of analgesics.

Mindfulness meditation requires the trainer to focus on breathing during the training process, while being non-critical and consciously observing various sensations on the body. It has a good effect in reducing pain, fatigue, negative emotions and strengthening coping with stressful events. With the rapid development of science and technology, meditation is no longer confined to traditional forms. The meditation method with the help of mobile communication technology and brain-computer interface technology can improve efficiency and convenience, and is more personalized. It has been recognized in many studies. The brain-computer interface is to establish a channel between the human brain and the computer that does not rely on conventional brain information output. Using techniques such as electroencephalogram, the spontaneous biopotential of the brain is amplified and recorded from the scalp.

This study aims to explore the impact of mindfulness meditation with devices based on brain-computer interface technology on patients undergoing radiofrequency ablation of atrial fibrillation. In order to improve the negative experience of patients during ablation, ensure the safety of patients during ablation, promote postoperative recovery, and increase satisfaction. The pain intensity, fatigue level, anxiety and depression of the meditation group and the control group were compared by the scale. Record relevant vital signs and adverse events.

The investigators hypothesized that the pain, fatigue, anxiety and depression of the meditation group would be lower than those of the control group.

DETAILED DESCRIPTION:
1. Research Background

   Atrial fibrillation is one of the most common arrhythmias in the world. According to 2020 ESC atrial fibrillation management guidelines, the global prevalence of atrial fibrillation is 2% to 4%. According to a 2021 epidemiological survey in china, there are about 7.9 million patients with atrial fibrillation in China over the age of 45. In the past 11 years, the prevalence of atrial fibrillation in China has increased 20-fold and has caused a huge financial and medical burden. In recent years, radiofrequency ablation has gradually become a first-line treatment for patients with atrial fibrillation. Radiofrequency ablation is an invasive procedure that lasts several hours, patients can experience varying degrees of discomfort and pain despite the use of analgesics. Studies have shown that more than 90% of patients have a strong sense of pain and discomfort during ablation even under deep sedation. In recent years, studies on mindfulness and meditation have been carried out among cardiac patients. Currently there is no application in radiofrequency ablation of atrial fibrillation. However, some studies have reported the application of visual hypnosis during atrial fibrillation ablation and turned out that it could help patients manage pain and anxiety. At the same time, patients have high treatment satisfaction. Studies have shown that meditation equipment based on brain-computer interface and artificial intelligence can show the state of the brain, help users conduct meditation training, and improve sleep. The application of such technologies in clinical nursing work provides new ideas.
2. Research purposes

   This study aims to explore the impact of mindfulness meditation with devices based on brain-computer interface technology on patients undergoing radiofrequency ablation of atrial fibrillation. In order to improve the negative experience of patients during surgery, ensure the safety of patients during surgery, promote postoperative recovery, and increase satisfaction. The pain intensity, fatigue level, anxiety and depression of the meditation group and the control group were compared by the scale. Record relevant vital signs and adverse events.
3. Research methods

   3.1.Sampling and grouping

   Use convenient sampling method to select patients and random number table grouping.

   3.2.Sample size calculation

   According to the calculation formula for comparing the two sample averages: n1= n2=2×(μα+μβ)2×σ2/δ2, where μα is the μ value of the first type of error probability (μ0.05=1.6449), and μβ is the second type The μ value of the error probability (μ0.10=1.2816), δ is the allowable error (the absolute value of the difference between the two groups of means), σ2=(Se2+Sc2)/2 (Se and Sc are respectively the study group and the control group Standard deviation). Substituting the above formula, calculating the sample size of each group of 36 cases, considering the 10% loss rate, the total number of cases is 80 cases.

   3.3.Ablation plan

   A unified ablation procedure was used. Analgesia plan: ①Parecoxib sodium 40mg + 10ml normal saline intravenous bolus; ②Fentanyl 0.4mg (4*2ml/piece) is configured to 40ml, fentanyl is initially 0.001mg/kg intravenously, and then the maintenance dose is 0.001mg /kg/h. If the patient complains of severe pain, speed up the analgesic bolus.

   3.4.Research team

   The research team includes 1 nursing management expert, 1 cardiologist, 2 clinical nurses, 1 clinical nurse who has obtained the national second-level psychological counselor certificate, and 1 nursing graduate student. Two nurses and two nursing graduate students were the main implementers of the intervention program. Psychology lecturers gave them a week of training in behavioral therapy and mindfulness meditation. All nurses in the cath lab have been trained by researchers and have mastered the methods of meditation training.
4. Outcome indicators

   4.1.normal information

   Gender, age, operation method, ablation time, number of discharges, energy, temperature, usage of anesthesia and analgesics, hypertension, diabetes, coronary heart disease, BMI, lvef, ladd, type of atrial fibrillation

   4.2.Specificity index

   Pain intensity, fatigue, anxiety and depression, heart rate, blood pressure, respiratory rate, pulse oxygen

   4.3.Adverse events
   1. The systolic blood pressure fluctuation is greater than 50mmHG
   2. Adverse drug reactions during surgery
   3. Vasovagal seizure
   4. Persistent chest pain between or after radiofrequency. Breathing disorders, such as difficulty breathing or shortness of breath.
5. Data collection method

Before intervention: collect general information and medical records

Intervention: Collect heart rate, blood pressure, pulse oxygen, number of patients reported pain, dosage of anesthesia and analgesics, duration of ablation, adverse events

After intervention: Collect pain score, anxiety and depression score

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Atrial Fibrillation
* Age ≥ 18 years
* First radiofrequency ablation treatment
* Informed consent, voluntary participation

Exclusion Criteria:

* With serious organic diseases such as malignant tumors
* With a history of mental illness or cognitive dysfunction, unable to correctly understand the questionnaire and intervention content
* Patients who are forced to or voluntarily withdraw due to changes in their condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Within 24 hours after radiofrequency ablation
  According to the International Pain Society, pain is an unpleasant subjective and emotional experience associated with existing or potential tissue damage and has been recognized as the fifth vital indicator. Using the Numeric Pain RatingScale(NPRS) to assess the patient's intraoperative pain level.0-10 means different degrees of pain, 0 means no pain, and 10 means the most severe pain. Patients choose the number that best represents their pain according to their own situation. 1-3 are mild pain, 4-6 are moderate pain, and 7-10 are severe pain.
the Brief Fatigue Inventory (BFI) | Within 24 hours after radiofrequency ablation
  Fatigue refers to continuous extreme exhaustion. The working ability, mental strength and physical strength are not as good as before. It is a subjective feeling, and this feeling cannot be relieved by rest. It is already a disease state or has become a factor in inducing other diseases. Using the Brief Fatigue Inventory(BFI) to assess the patient's fatigue. According to the presence or absence of fatigue symptoms, it is represented by 0-10, 0 means no fatigue, and 10 means severe fatigue that cannot be relieved.
the State-trait anxiety inventory (STAI) | Within 24 hours after radiofrequency ablation
  Use the (STAI, Form YI) part of the State-trait anxiety inventory (STAI) to assess anxiety. This scale is mainly used to assess the immediate or recent experiences or feelings of fear, tension, anxiety and neuroticism at a specific time or situation .

SECONDARY OUTCOMES:
heart rate | pre ablation, 10 minutes after ablation begin, 20 minutes after ablation begin, 30 minutes after ablation begin, 10minutes after ablation
  Heart rate refers to the number of heartbeats per minute of normal people in a quiet state, also called resting heart rate, generally 60-100 beats/min. An ECG monitor is used for continuous monitoring. The heart rate will increase under stressful conditions such as tension and pain.
blood pressure | pre ablation, 10 minutes after ablation begin, 20 minutes after ablation begin, 30 minutes after ablation begin, 10minutes after ablation
  Blood pressure refers to the lateral pressure acting on the blood vessel wall per unit area when the blood flows in the blood vessel, and it is the driving force to promote the blood flow in the blood vessel. An electronic sphygmomanometer is used for monitoring. The blood pressure range of normal adults in a quiet state is relatively stable, with a normal range of systolic blood pressure of 90～139mmHg, diastolic blood pressure of 60～89mmHg, and pulse pressure of 30～40mmHg.
respiratory rate | pre ablation, 10 minutes after ablation begin, 20 minutes after ablation begin, 30 minutes after ablation begin, 10minutes after ablation
  Adopting the breathing monitoring function of the ECG monitor, the normal adult breathing rate is 12-20 times per minute.
pulse oxygen | pre ablation, 10 minutes after ablation begin, 20 minutes after ablation begin, 30 minutes after ablation begin, 10minutes after ablation
  Pulse oxygen refers to the blood oxygen saturation detected by the device at the end of the hand, which can indirectly reflect whether the body is hypoxic. The normal level is greater than 94%.

OTHER OUTCOMES:
intraoperative adverse reaction | intraoperative (during the operation)
  excessive blood pressure fluctuations (systolic blood pressure fluctuations greater than 50mmHG), intraoperative drug adverse reactions (such as nausea and vomiting), vasovagal reaction, persistent chest pain during or after ablation
number of oral reports of pain during surgery | intraoperative (during the operation)
  Record the number of spontaneous oral complaints of pain during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhipeng Bao, Master, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] He Y, Tang Z, Sun G, Cai C, Wang Y, Yang G, Bao Z. Effectiveness of a Mindfulness Meditation App Based on an Electroencephalography-Based Brain-Computer Interface in Radiofrequency Catheter Ablation for Patients With Atrial Fibrillation: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 May 3;11:e44855. doi: 10.2196/44855. PMID 37133926